CLINICAL TRIAL: NCT01576120
Title: Evaluation of a PillCam Colon Bowel Preparation Regimen in Crohn's Disease Patients- Pivotal Study
Brief Title: Evaluation of a PillCam Colon Bowel Preparation Regimen in Crohn's Disease Patients
Acronym: RD-207
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RD-207
Record Dates: First submitted 2012-04-05; First posted 2012-04-12 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2014-10

CONDITIONS: Crohn's Disease
Keywords: Known, active Crohn's disease; Iieocolonic or colonic involvement; proven patency of the GI tract
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bowel prep regimen first boost 6 oz. and second boost 3 oz. (Experimental): 4L of PEG split into two doses:1.on the evening before the exam 2.on the morning of exam day.Upon SB Detection 6 oz. SuPrep administered and 3hrs later 3 oz. SuPrep was administered if needed depends on the capsule progress in the GI
  Interventions: Other: bowel prep regimen first boost 6 oz. and second boost 3 oz.
- bowel prep regimen first boost 3 oz. and second boost 6 oz. (Experimental): 4L of PEG split into two doses:1.on the evening before the exam 2.on the morning of exam day.Upon SB Detection 3 oz. SuPrep administered and 3hrs later 6 oz. SuPrep was administered if needed depends on the capsule progress in the GI
  Interventions: Other: bowel prep regimen first boost 3 oz. and second boost 6 oz.

INTERVENTIONS:
Other: bowel prep regimen first boost 6 oz. and second boost 3 oz. — Subjects will be instructed to perform the bowel preparation procedure and follow a detailed dietary regimen prior to and during the CE procedure.
  In this arm the subjects administered a 6 oz. dose of Suprep as first boost and if needed addtional 3 oz. of Suprep (second boost)
  Arms: bowel prep regimen first boost 6 oz. and second boost 3 oz.
Other: bowel prep regimen first boost 3 oz. and second boost 6 oz. — Subjects will be instructed to perform the bowel preparation procedure and follow a detailed dietary regimen prior to and during the CE procedure.
  In this arm the subjects administered a 3 oz. dose of Suprep as first boost and if needed addtional 6 oz. of Suprep (second boost)
  Arms: bowel prep regimen first boost 3 oz. and second boost 6 oz.

SUMMARY:
The proposed study is designed to evaluate Pillcam regimen in Crohn's disease patients, using the PillCam Colon system.

DETAILED DESCRIPTION:
1. Primary Scientific Objective Evaluate the effectiveness of the PillCam COLON 2 Prep Regimen in CD patients.

   Secondary Objective To evaluate safety of the PillCam™ COLON 2 procedure in CD patients
2. Study Hypothesis Crohn's Disease may be pan-enteric in nature and can affect the small bowel, the colon or both. PillCam COLON 2 may be used for visualization of both SB and colon mucosa in Crohn's Disease patients. However, bowel prep is required in order to evacuate all fecal matter prior to the exam and in order to propel the capsule and complete its traverse through the entire GI track within examination time.
3. The study is designed to evaluate the effectiveness of the prep regimen in terms of transit, excretion and cleansing in CD patients

All end points will be evaluated within 4 months from end of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age and above

  * Subjects who are determined by their physician to have active Crohn's disease based on at least one of the following tests which were performed in the past 3 months :

    * Colonoscopy
    * Capsule endoscopy of the small bowel or colon
    * Other radiology tests
    * Clinical symptoms with elevated positive inflammatory markers ;ESR, CRP, thrombocytosis, leukocytosis, fecal lactoferrin, or fecal alpha-1 antitrypsin
  * Proven patency by the Agile capsule or another approach deemed clinically acceptable by the investigator, e.g. CT enterography, performed within the 3 months prior to enrollment
  * Subject is able and agrees to sign the Informed Consent Form

Exclusion Criteria:

* • Subject has dysphagia

  * Subject has congestive heart failure
  * Subject has renal insufficiency
  * Subject has cirrhosis
  * Subject is known or is suspected to suffer from intestinal obstruction
  * Subject has known previous stricture/obstruction of the SB or colon
  * Chronic use of laxatives
  * Subject has a cardiac pacemaker or other implanted electro medical device.
  * Women who are either pregnant or nursing at the time of screening, who intend to be during the study period, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
  * Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
  * Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator.
  * Subject has any condition, which precludes compliance with study and/or device instructions.
  * Subject suffers from life threatening conditions
  * Subject is currently participating in another clinical study
  * Subject has known slow gastric emptying time or GI transit time.
  * Subject is allergic or contraindicated to any of the study medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Dayton Gastroenterology, Beavercreek, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Bowel Prep Regimen First Boost 6 oz. and Second Boost 3 oz.: 4L of PEG split into two doses:1.on the evening before the exam 2.on the morning of exam day.Upon SB Detection 6 oz. SuPrep administered and 3hrs later 3 oz. SuPrep was administered if needed depends on the capsule progress in the GI
  bowel prep regimen first boost 6 oz. and second boost 3 oz.: Subjects will be instructed to perform the bowel preparation procedure and follow a detailed dietary regimen prior to and during the CE procedure.
  In this arm the subjects administered a 6 oz. dose of Suprep as first boost and if needed addtional 3 oz. of Suprep (second boost)
- Bowel Prep Regimen First Boost 3 oz. and Second Boost 6 oz.: 4L of PEG split into two doses:1.on the evening before the exam 2.on the morning of exam day.Upon SB Detection 3 oz. SuPrep administered and 3hrs later 6 oz. SuPrep was administered if needed depends on the capsule progress in the GI
  bowel prep regimen first boost 3 oz. and second boost 6 oz.: Subjects will be instructed to perform the bowel preparation procedure and follow a detailed dietary regimen prior to and during the CE procedure.
  In this arm the subjects administered a 3 oz. dose of Suprep as first boost and if needed addtional 6 oz. of Suprep (second boost)
Period: Overall Study
Arm/Group | Bowel Prep Regimen First Boost 6 oz. and Second Boost 3 oz. | Bowel Prep Regimen First Boost 3 oz. and Second Boost 6 oz.
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bowel Prep Regimen First Boost 6 oz. and Second Boost 3 oz. | Bowel Prep Regimen First Boost 3 oz. and Second Boost 6 oz. | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (10.9) | 39.7 (11.7) | 37.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: • Evaluate the Effectiveness of the PillCam COLON 2 Bowel Prep Regimen in Crohn's Disease Patients
Description: effectiveness of the PillCam COLON 2 bowel prep regimen in Crohn's Disease patients will be evaluated by the folloiwng: • Bowel preparation cleansing level assessment
  The duration of the procedure in this study is 1 day of colon preparation and
  1 day of Capsule Endoscopy (CE) procedure. 5-9 days after the CE procedure a follow up call to the subjects will be conducted.
Time Frame: The end points and outcomes measures will be evaluated within 4 months from end of enrollment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bowel Prep Regimen First Boost 6 oz. and Second Boost 3 oz. | Bowel Prep Regimen First Boost 3 oz. and Second Boost 6 oz.
Number analyzed (Participants) | 21 | 19
percentage of participants | 62 [38 to 62] | 79 [54 to 94]

ADVERSE EVENTS:
Arm/Group | Bowel Prep Regimen First Boost 6 oz. and Second Boost 3 oz. | Bowel Prep Regimen First Boost 3 oz. and Second Boost 6 oz.
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 9/21 | 4/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bowel Prep Regimen First Boost 6 oz. and Second Boost 3 oz. (N=21) | Bowel Prep Regimen First Boost 3 oz. and Second Boost 6 oz. (N=19)
Adverse event related to the preparation (Gastrointestinal disorders) | 6 | 2 — adverse events were reported as related to the the preparation such as vomiting and nausea
Adverse event not related to study procedure (Gastrointestinal disorders) | 3 | 2 — adverse events were reported as not related to the study procedure such as fever and headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No